CLINICAL TRIAL: NCT00646958
Title: A Phase 2, Multicenter, Randomized, Open-Label, Comparative Study to Evaluate the Safety and Efficacy of RX-1741 Versus Linezolid in the Outpatient Treatment of Adult Patients With Uncomplicated Skin and Skin Structure Infection
Brief Title: Safety and Efficacy Study of Oxazolidinones to Treat Uncomplicated Skin Infections
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Melinta Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RX-1741-202
Record Dates: First submitted 2008-03-26; First posted 2008-03-31 (Estimated); Results first posted 2009-06-26 (Estimated); Last update posted 2014-03-27 (Estimated); Status verified 2014-02

CONDITIONS: Infectious Skin Diseases; Bacterial Skin Diseases; Staphylococcal Skin Infections; Streptococcal Infections; Abscess
MeSH Terms: conditions — Skin Diseases, Infectious; Skin Diseases, Bacterial; Staphylococcal Skin Infections; Streptococcal Infections; Abscess | interventions — radezolid; Linezolid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Radezolid 450 mg PO QD
  Interventions: Drug: Radezolid
- 2 (Experimental): Radezolid 450 mg PO BID
  Interventions: Drug: Radezolid
- 3 (Active Comparator): Linezolid 600 mg PO BID
  Interventions: Drug: Linezolid

INTERVENTIONS:
Drug: Radezolid — 450mg PO QD
  Other Names: RX-1741
  Arms: 1
Drug: Radezolid — 450mg PO BID
  Other Names: RX-1741
  Arms: 2
Drug: Linezolid — 600mg PO BID
  Other Names: Zyvox
  Arms: 3

SUMMARY:
The purpose of this study is to assess the efficacy, safety and tolerability of RX-1741, an oxazolidinone, versus linezolid, another oxazolidinone, in the treatment of uncomplicated skin and skin structure infections

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with uSSSI
* Adult (men and women) ≥18 years
* Females must be post-menopausal for at least 1 year or surgically sterile
* Sexually active males must use a barrier method of birth control during and for 30 days after the study
* Acceptable clinical diagnoses of uSSSI include, but are not limited to: Simple abscess, Impetiginous lesions, Folliculitis, Furunculosis, Carbuncles, Cellulitis
* The infection is accompanied by 2 or more of the following local signs and symptoms: Pain/tenderness, Swelling, Erythema, Localized warmth, Purulent drainage/discharge, Induration, Regional lymph node swelling or tenderness, Extension of redness
* A sample for microbiologic culture must be obtained from the primary infection site at the screening visit
* The patient must require and be a suitable candidate for oral antibiotic therapy in the opinion of the Investigator and be able to swallow tablets or capsules intact
* A written, voluntarily signed informed consent must be obtained from the patient prior to the initiation of any study-related procedures

Exclusion Criteria:

* Cellulitis (area greater than 10cm2), chronic or recurrent furunculosis, postoperative wound infection, leg ulcer, decubitus ulcer(s), erysipelas, progressive lymphangitis, acute paronychia or a deep tissue abscess such as pilonidal or breast abscess. Also excluded are skin infections resulting from animal bites
* Patients with a complicated skin and skin structure infection as judged by the Investigator
* Infections that can be treated by surgical incision alone according to the judgment of the Investigator
* Treatment with the following anti-infective agents prior to study drug administration: systemic antibiotic within 7 days; azithromycin within 14 days; a long-acting injectable antibiotic within 30 days
* Any infection which requires the use of a concomitant antimicrobial agent, in addition to study drug
* Concomitant topical therapy at the infection site for the period within 48 hours prior to study drug administration through TOC
* A chronic or underlying skin condition at the site of infection or infections involving prosthetic materials
* A wound secondary to burn injury or acne vulgaris
* Any infection site that requires: intraoperative surgical debridement; excision of infected area
* Documented or suspected bacteremia
* Fungal infection involving the nail bed or scalp at the primary uSSSI site
* Significant peripheral vascular disease
* An abscess at an anatomical location where the incidence of anaerobic pathogen involvement is increased
* Patient receiving a daily dose of > 15 mg of systemic prednisone or equivalent, for > 10 days within the period starting 14 days prior to study drug administration or anticipated through TOC
* Patient with known human immunodeficiency virus (HIV) infection.
* Medical history of hypersensitivity or allergic reaction to linezolid according to the judgment of the Investigator
* Patients receiving serotonergic agents, selective serotonin reuptake inhibitors (SSRIs), or monoamine oxidase inhibitors (MAOIs)
* Patients who have severe liver disease
* History of pheochromocytoma, untreated hyperthyroidism, untreated or uncontrolled hypertension, carcinoid syndrome
* Evidence of uncontrolled, clinically significant (according to the judgment of the Investigator) cardiovascular, pulmonary, metabolic, gastrointestinal, neurological, or endocrine disease; malignancy or psychiatric disorder
* Current evidence of deep vein thrombosis or superficial thrombophlebitis
* Experienced a recent clinically significant coagulopathy
* Evidence of clinically significant immunosuppression
* Patient who previously enrolled in this study
* Patient who has previously enrolled in any other clinical trial within 4 weeks of enrollment through TOC. Treatment with an investigational drug within 4 weeks prior to study drug administration
* Patient residing in a chronic care facility
* Any underlying condition or disease state that would interfere with the completion of the study procedures and evaluation of the absorption of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2007-12; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Hopkins, MD, Study Director — Melinta Therapeutics, Inc.
Locations (19):
- United States (19):
  - Drug Research & Analysis Corp, Montgomery, Alabama
  - OWENS Pharma Research Center, Long Beach, California
  - Healthcare Partners Medical Group, Los Angeles, California
  - HealthCare Partners Medical Group, Pasadena, California
  - Olive View- UCLA Center, Dept. Emergency Medicine, Sylmar, California
  - South Florida Clinical Research, Atlantis, Florida
  - Southeast Regional Research Group, Columbus, Georgia
  - Contemporary Medicine, LLC, Hinesville, Georgia
  - Infectious Disease of Indiana, PSC., Indianapolis, Indiana
  - Clinical Trials of America, Inc., Shreveport, Louisiana
  - Arnold Markowitz, MD., PC, Keego Harbor, Michigan
  - Mercury Street Medical Group, LLC, Butte, Montana
  - Jamaica Hospital Medical Center, Jamaica, New York
  - ALL-TRIALS Clinical Research, LLC, Winston-Salem, North Carolina
  - Summa Health System, Akron, Ohio
  - Brandywine Clinical Research, Downington, Pennsylvania
  - Warminster Medical Associates, P.C., Warminster, Pennsylvania
  - McKenzie Medical Center, McKenzie, Tennessee
  - J. Lewis Research, Inc., Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study targeted participants with uncomplicated skin and soft tissue infections (uSSSI) for which oral, outpatient treatment was appropriate. Eligible uSSSIs included simple abscesses, impetigo, folliculitis, furunculosis, carbuncles, and cellulitis (area <10 cm2).
Groups:
- Radezolid QD: 450 mg by mouth (PO) once daily (QD)
- Radezolid BID: 450 mg by mouth (PO) twice daily (BID)
- Linezolid BID: 600 mg by mouth (PO) BID
Period: Overall Study
Arm/Group | Radezolid QD | Radezolid BID | Linezolid BID
Started | 51 (Number (No.) Participants Randomized) | 50 (No. Participants Randomized) | 49 (No. Participants Randomized)
Completed | 40 | 41 | 40
Not Completed | 11 | 9 | 9
Not completed — Lack of Efficacy | 1 | 0 | 0
Not completed — Adverse Event | 4 | 0 | 0
Not completed — Lost to Follow-up | 1 | 5 | 7
Not completed — Protocol Violation | 1 | 1 | 0
Not completed — Abnormal screening lab tests | 1 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 0
Not completed — Did not receive study drug | 2 | 0 | 2

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) population included those patients who were randomized and took at least one (1) dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Radezolid QD | Radezolid BID | Linezolid BID | Total
Number analyzed (Participants) | 51 | 50 | 49 | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.8 (12.43) | 43.6 (13.65) | 43.7 (16.33) | 43.3 (14.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 14 | 13 | 41
  Male | 37 | 36 | 36 | 109

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Clinical Response of Cure
Description: To qualify as a Cure, participants were required to fulfill the following criteria: all systemic signs and symptoms of uSSSI present at screening were improved or resolved; no further antibiotic therapy was necessary for treatment of uSSSI; and there was no worsening or appearance of new signs and symptoms of uSSSI.
Time Frame: Test of Cure (TOC), day 10-20
Population: Clinically Evaluable participants were those that met the entry criteria, received a certain amount of drug, did not receive any additional antibiotics before Test of Cure (TOC), and who presented for a TOC evaluation in the appropriate window.
Measure: Number; unit: Participants
Arm/Group | Radezolid QD | Radezolid BID | Linezolid BID
Number analyzed (Participants) | 39 | 36 | 38
Participants | 38 | 34 | 37

2. Secondary Outcome: Number of Patients With Per-Patient Microbiologic Response of Eradicated
Description: The microbiological response at the patient level was considered Eradicated (documented or presumed)if no pathogens were present in repeat cultures taken from the original site of infection or a clinical response of cure precluded the ability to obtain a culturable specimen.
Time Frame: Test of Cure (TOC), day 10-20
Population: Microbiologically Evaluable patients were those that met the entry criteria, received a certain amount of drug, did not receive any additional antibiotics before TOC, presented for a TOC evaluation in the appropriate window, and who had a baseline pathogen that was susceptible to study drug.
Measure: Number; unit: Participants
Arm/Group | Radezolid QD | Radezolid BID | Linezolid BID
Number analyzed (Participants) | 20 | 26 | 23
Participants | 20 | 23 | 21

ADVERSE EVENTS:
Time Frame: Safety was monitored as follows: on Day 1 (after signing the informed consent), and on Days 5 (on therapy) +/-1; 5-10 (EOT) +/-1; and 10-20 (TOC) +/-1. All SAEs and any AEs ongoing at TOC were followed until they either resolved or were deemed stable.
Description: While 51, 50 and 49 subjects were randomized to radezolid qd, radezolid bid, and linezolid, respectively, safety was assessed in the ITT population (those who received at least 1 dose of study drug.) Four subjects (2 in radezolid qd and 2 in linezolid) did not receive any study drug; thus, the # of subjects at risk is 49, 50 and 47, respectively.
Arm/Group | Radezolid QD | Radezolid BID | Linezolid BID
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/50 | 0/47
Other Adverse Events (participants affected / at risk) | 20/49 | 17/50 | 10/47
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Radezolid QD (N=49) | Radezolid BID (N=50) | Linezolid BID (N=47)
Diarrhea (Gastrointestinal disorders) | 11 | 11 | 1
Headache (Nervous system disorders) | 6 | 3 | 3
Nausea (Gastrointestinal disorders) | 4 | 1 | 3
Elevated AST (Investigations) | 2 | 0 | 0
Abnormal LFT (Investigations) | 0 | 2 | 1
Somnolence (Nervous system disorders) | 0 | 2 | 0
Infections and infestations (Infections and infestations) | 2 | 0 | 0
Investigations (Investigations) | 3 | 4 | 4

LIMITATIONS AND CAVEATS:
This was an unblinded study, which raises the possibility of bias.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor retains control of all publication rights.